CLINICAL TRIAL: NCT07050979
Title: Goal-Directed Fluid Therapy Versus Conventional Fluid Therapy for Thoracoscopic Lobectomy in the ERAS Era: A Randomized Controlled Trial
Brief Title: Goal-Directed Fluid Therapy for Thoracoscopic Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Demet Laflı Tunay, Associate Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GDFTinERAS
Record Dates: First submitted 2025-06-23; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Thoracoscopic Lobectomy; Thoracic Anesthesia; Enhanced Recovery After Anesthesia; Lung Cancer
Keywords: Goal directed fluid therapy; Enhanced Recovery After Anesthesia; Pressure Recording Analytical Method; Stroke volume variation; Cardiac index
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients meeting the inclusion criteria were randomized into the intervention (goal directed fluid therapy - group GDFT, n=40) or control (conventional fluid therapy - control group, n=40) groups using opaque sealed envelopes.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist responsible for intraoperative management was aware of the group assignments, but other members of the research team, other healthcare providers, and patients were unaware. Confidentiality of randomization to the investigators was maintained until the end of the study for statistical data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-Directed Fluid Therapy (GDFT) (Experimental): Patients receive intraoperative fluid and vasopressor therapy guided by Stroke Volume Variation (SVV < 15%) and Cardiac Index (CI > 2.6 L/min/m²) using the Pressure Recording Analytical Method (PRAM). Basal fluid replacement is provided with 5 mL/kg/hour Lactated Ringer's solution.
  Interventions: Other: Goal-Directed Fluid Therapy (GDFT)
- Conventional Fluid Therapy (Active Comparator): Patients receive intraoperative fluid and vasopressor therapy targeting Mean Arterial Pressure (MAP) of 65-95 mmHg and minimum hourly urine output of 0.5 mL/kg/hour. Basal fluid replacement is provided with 5 mL/kg/hour Lactated Ringer's solution.
  Interventions: Other: Conventional Fluid Therapy

INTERVENTIONS:
Other: Goal-Directed Fluid Therapy (GDFT) — This arm administers fluid and vasopressor therapy based on SVV (less than 15%) and CI (>2.6 L/min/m²) targets using the Pressure Recording Analytical Method (PRAM) system with the help of intra-arterial pressure monitoring method. Basal fluid replacement is provided with 5 mL/kg/hr of Lactated Ringer's solution.
  Arms: Goal-Directed Fluid Therapy (GDFT)
Other: Conventional Fluid Therapy — This arm administers fluid and vasopressor therapy based on targets of Mean Arterial Pressure (MAP) 65-95 mmHg and hourly urine output minimum of 0.5 mL/kg/hr. Basal fluid replacement is provided with 5 mL/kg/hr of Lactated Ringer's solution.
  Arms: Conventional Fluid Therapy

SUMMARY:
The investigators aimed to examine the effect of goal-directed fluid therapy (GDFT) compared to conventional fluid therapy in thoracoscopic lobectomy surgery with ERAS protocol on intraoperative pulmonary oxygenation and 30-day patient outcomes including postoperative morbidity and mortality. The primary outcome measure of the study was the PaO2/FiO2 ratio (change in pulmonary oxygenation) during one-lung ventilation, and the secondary outcomes were postoperative morbidity, quality of recovery, 30-day re-admission, and mortality rate.

This randomized controlled study analyzed 80 adult patients who underwent thoracoscopic lobectomy surgery with the ERAS protocol. In addition to standard monitoring in the operating room, all participants underwent Pressure Recording Analytical Method (PRAM) monitoring with the help of intra-arterial pressure monitoring method. Participants were randomly assigned to GDFT and conventional fluid therapy groups. In the GDFT group, fluid, inotropic agent and/or vasopressor therapy was administered by targeting stroke volume variation (SVV) and cardiac index (CI). In the control group, fluid and/or vasopressor therapy was administered with the guidance of MAP 65-95 mmHg and urine output at least 0.5 mL/kg/hr. Intraoperative hemodynamic data, amount and types of fluid administered, inotropic and vasopressor agents were recorded. Vital signs, pulmonary, cardiac and other system morbidity, quality of recovery on days 1, 3 and 5 in the postoperative care unit and in the ward, and re-admission to hospital and mortality within 30 days were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* ASA Physical Status Classification I-II.
* Undergoing elective thoracoscopic lobectomy with the ERAS protocol.
* Provided informed consent.

Exclusion Criteria:

* Age < 18 or > 65 years.
* ASA Physical Status Classification III or higher.
* Patients not in sinus rhythm, and with recent oral beta-blocker use.
* Patients with cardiac/renal/hepatic insufficiency, valvular heart disease (aortic or mitral valve insufficiency or stenosis)
* Patients with abnormal preoperative lung function (forced expiratory volume in 1 second less than 50% of predicted values)
* Patients with severe obesity (BMI>35 kg/m2)
* Patients who cannot be applied to the ERAS protocol
* Emergency surgery.
* Refusal to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Change in PaO2/FiO2 Ratio During One-Lung Ventilation | Intraoperative period (from anesthesia induction to extubation).
  Measurement of PaO2/FiO2 ratio at five time points intraoperatively to assess pulmonary oxygenation.

SECONDARY OUTCOMES:
Postoperative Pulmonary Complications | Up to postoperative day 5.
  Incidence of pulmonary complications (e.g., pulmonary edema, atelectasis, acute lung injury) assessed using chest X-ray and clinical evaluation.
Postoperative Cardiac Complications | Up to postoperative day 5.
  Incidence of cardiac complications (e.g., hypotension, hypertension, dysrhythmia).
Postoperative Renal Complications | Up to postoperative day 5.
  Incidence of acute kidney injury (AKI).
Postoperative Infectious Complications | Up to postoperative day 5.
  Incidence of infections (e.g., pneumonia, surgical site infection).
Quality of Recovery (QoR-15 Score) | Postoperative 24th hour.
  Patient-reported recovery quality assessed using the QoR-15 scale.
Length of Hospital Stay | From date of surgery until the date of discharge.
  Duration of hospital stay in days.
30-Day Hospital Readmission Rate | From date of discharge until the postoperative 30th day.
  Rate of hospital readmissions within 30 days post-surgery.
Mortality Rate | Postoperative 30th day.
  Incidence of mortality within 30 days post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Saricam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided